CLINICAL TRIAL: NCT05639101
Title: GeoAsma: Pilot and Evaluation of a Clinical Decision Support System and a Mobile App for the Management of Asthma Patients.
Acronym: GeoAsma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Principal Investigator, Alberto Moreno Conde, PHD Alberto Moreno Conde, Hospital Universitario Virgen Macarena
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI-0100-2020
Record Dates: First submitted 2022-08-01; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Decision support system for professionals and mobile app for self-management in patients based on the analysis of the influence of clinical and environmental characteristics on the population of asthmatic patients in our region.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Clinicians will use a Clinical decision support system to better manage their patients. Asthmatic patients will use a smartphone app for their self management.
  Interventions: Other: Clinical Decission support system management & mobile App Intervention Group
- Control (No Intervention): Asthmatic patients that will not be subject to any intervention

INTERVENTIONS:
Other: Clinical Decission support system management & mobile App Intervention Group — The clinicians treating the patients will use a clinical decision support system that includes predictive models associated with the level of risk of exacerbation. This models have been obtained in asthmatic patients by applying data mining techniques and multilevel analysis in the study of the influence of clinical characteristics and the environment of each subject.
  The patients will use a mobile app to help manage their symptoms.
  Arms: Intervention group

SUMMARY:
GeoAsma is a study for the definition, validation and evaluation of predictive models on the influence of the environment on asthmatic patients in Andalusia.

DETAILED DESCRIPTION:
Although for decades there have been multiple studies on the association of asthma with factors such as weather conditions, pollution, pollen and the social condition of patients, the GeoAsma project aims to advance the study of environmental factors that influence the health of asthmatic patients by combining BigData technology and data mining analysis, Geographic Information Systems and open data provided by official sources with data from the Electronic Health Record of the Andalusian Health System, that provides healthcare services to more than 8,000,000 citizens.

This project aims to study through data mining techniques and multilevel analysis the influence of clinical and environmental factors: pollen level, air pollution, atmospheric conditions and social determinants in more than 800,000 asthmatic patients during the last 15 years in Andalusia, the southernmost region of Spain. It is expected that the results of this study will serve to define predictive models that will help professionals and patients in our region to make decisions.

After the validation of the models, a decision support system will be implemented in a web platform and in a mobile application. Its impact on the reduction of exacerbations, control, quality of life and resource consumption of asthmatic patients will be analysed. This evaluation will be carried out through a pilot with 214 patients with a follow-up period of 12 months with asthma in the hospitals participating in this proposal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bronchial asthma in its intermittent and persistent degrees mild/moderate.
* No respiratory infections in the month prior to testing.
* Availability and/or ability to use a Smartphone.

Exclusion Criteria:

* Severe persistent asthmatics.
* Pregnant women, breastfeeding women or women who want to become pregnant during the duration of the study.
* Subjects with malignant disease, uncontrolled risk factors or any pathology that compromises the safety of the study.
* Treatment with systemic corticosteroids during the 6 months prior to or during the study.
* Subjects with problems that limit their ability to cooperate.
* Subjects unable to perform correct spirometric maneuvers.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Asthma control | 1 year
  The Asthma Control Test is a validated determination of asthma control that is directly control of asthma that is answered directly by the patient and consists of five questions questions that assess: activity limitations, dyspnea, nocturnal symptoms, rescue medication use, and the patient's overall rating of asthma control. symptoms, use of rescue medication, and the patient's overall rating of asthma control over the previous four weeks, which is defined from the results of a questionnaire.
Number of exacerbations Number of exacerbations | 1 year
  Measured by the number of times the patient goes to the emergency room or uses rescue medication and/or cycles of oral corticosteroids.
Health-related quality of life | 1 year
  The Asthma Quality of Life Questionnaire (AQLQ) will be administered at baseline, 3 and 6 months of the study. The AQLQ contains 32 items corresponding to 4 dimensions of health: limitation of usual activities, symptoms, emotional function, and environmental stimuli.
Quality-adjusted life year | 1 year
  To calculate this index, the EuroQol-5D quality of life questionnaire will be administered at baseline, three and six months into the study. The EQ-5D describes health status with five dimensions (mobility, self-care, activities of daily living, pain/discomfort, and anxiety/depression), each of which is defined with three levels of severity. It also consists of a millimetered Visual Analog Scale (VAS) on which the subject must score his or her health status on the day of the survey, with the extremes of the scale being the worst imaginable health status (0) and the best imaginable health status (100).
Patient satisfaction | 1 year
  It will be carried out at the end of the study by means of a questionnaire that includes items on ease of use, usefulness, intention to use, etc.
Respiratory function | 1 year
  Several pulmonary function tests will be carried out. These tests will include spirometry (FEV1, FVC, FEV1/FVC ratio, PC20, PD15, Fractional exhaled nitric oxide)
Immune response | 1 year
  IgE test, lymphocite count
Treatment adherence | 1 year
  Estimated through dispensations

SECONDARY OUTCOMES:
Economic evaluation | 1 year
  Incremental cost-efectiveness ratio and incremental cost-utility ratio between the intervention group and control group

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Moreno, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Alberto Moreno Conde, Seville, Spain

IPD SHARING:
Plan to Share IPD: No